CLINICAL TRIAL: NCT01850199
Title: Intelligent and Educational System for Gestational Diabetes Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: CIBER-BBN: Networking Research Center for Bioengineering. (Unknown); Technical University of Madrid (Other)
Responsible Party: Principal Investigator, Mercedes Rigla, Director, Endocrinology and Nutrition Dpt., Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SINEDiE
Record Dates: First submitted 2013-05-03; First posted 2013-05-09 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Gestational Diabetes
Keywords: Gestational diabetes; Telemedicine; Artificial Intelligence
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual management (presential visits) (Active Comparator): Patient will follow the usual care program, which includes in-person appointment (weekly/biweekly)
  Interventions: Other: Usual management
- Smart telemedicine remote monitoring for gestational diabetes (Experimental): After receiving an structured education on the matter, patients will be followed remotely by analysing glucose and diet/physical activity/other events data with a periodicity no longer than 48 hours
  Interventions: Other: Smart telemedicine remote monitoring for gestational diabetes

INTERVENTIONS:
Other: Smart telemedicine remote monitoring for gestational diabetes — Intervention consists of a telemedicine platform which includes artificial intelligence tools to analyse glucose values and guarantee an optimal glucose control from the diagnosis of gestational diabetes to delivery.
  Arms: Smart telemedicine remote monitoring for gestational diabetes
Other: Usual management — Usual care will be provided, including face-to-face visits
  Arms: Usual management (presential visits)

SUMMARY:
Gestational diabetes, diabetes diagnosed during pregnancy, affects 8.8% of pregnancies in Spain that means more than 40,000 women per year. This prevalence is based on the National Diabetes Data Group criteria, previous to the 4th workshop on Gestational Diabetes (1998), but, if the new diagnosis criteria proposed by the International Associations of Diabetes and Pregnancy Study Groups, based on the most important study never made before on this topic, prevalence would increase to the double. When a women is diagnosed, the risk of complications for her and the child increases and, therefore, she has to start an specific diet and frequent visits to the diabetes center in order to check that glucose values do not exceed 95 mg/dl before or 140 mg/dl 1-hour after meals. In other case, she should start insulin treatment. Our project is aimed to develop intelligent tools based on neuro-diffuse techniques and integrated in a telemedicine system that allows control of gestational diabetes automatically, guaranteeing glucose control objectives consecution and avoiding face-to-face visits to the health care center. Furthermore, educational and motivation tools for a healthy behaviour will be included. At the end of the study efficacy and security about insulin management will be compare with the recommendations proposed by the diabetes team and data about direct and indirect costs will be calculated. The investigators anticipate that the smart telemedicine system can allow us to detect high blood glucose values earlier than in-person scheduled visits.

DETAILED DESCRIPTION:
This study aims to evaluate the safety and usability of a telemedicine system which includes intelligent tools for blood glucose analysis and supporting routine clinical monitoring carried out by nurses and endocrinologists.

Type of study: Prospective, controlled, randomized (2:1) Participants: pregnant women diagnosed with gestational diabetes according to the National Diabetes Data Group criteria between 14 and 34 weeks of gestation. Patients with suspected clinical diagnosis of type 1 or type 2 diabetes will be excluded.

In addition to the signed acceptance to participate in the study, requirements are:

* Availability of a desktop computer or laptop with an internet connection and USB port.
* Sufficient knowledge of Catalan and/or Spanish
* A mobile phone Objective: To technically evaluate the SineDie telemedicine system and also the users' degree of satisfaction.

Methodology of the study: Once signed consent for participation the patient will be randomized either to continue regularly scheduled visits (33% chance) or to use the Telemedicine system (66% chance). The randomization will be done using a system of allocation based on random numbers. The SINEDiE system includes:

* Educational Program
* Automatical Evaluation of glucose data -immediately after each download (frequency not exceeding 72 hours)
* Alerts in case of failure of receiving information at the scheduled time or in case of incompleteness.
* Alerts for glucose values higher than desirable but which could be corrected by diet changes and / or exercise
* Alerts for high glucose values which cannot be corrected with the previous mentioned changes. In this case an appointment for face-to-face visit would be made.

All warnings are also reported as an email to the endocrinologist and nurse

Variables:

* Statistical analysis of data: blood glucose, standard deviation, number of preprandial values> 90, the number of postprandial values of> 140 messages and warnings
* Analytical variables: HbA1c at the start and every 4 weeks
* Complications of pregnancy and childbirth if any.
* Neonatal Complications if any
* Survey of satisfaction with telemedicine tool

Expected duration of the study: 6 months Number of patients included 20 patients

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy; Gestational diabetes diagnosed according the National Diabetes data Group Criteria.

Exclusion Criteria:

* Pregestational diabetes (diagnosed or suspected); Illiteracy; no computer connected to internet availability; unwillingness to participate in the study

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Median blood glucose (Interquartile range) | From inclusion to delivery (estimate average period 10±2 weeks)
  Blood glucose data downloaded from the glucometer will allow to obtain the main outcome.

SECONDARY OUTCOMES:
Time from glucose criteria for insulin prescription to actual insulin starting | From inclusion to delivery From inclusion to delivery (estimate average period 10±2 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Parc Tauli Sabadell University Hospital, Sabadell, Barcelona, Spain